CLINICAL TRIAL: NCT03568630
Title: A Longitudinal Cohort Study to Identify Clinical and Blood Markers of Early Pancreas Cancer
Brief Title: Blood Markers of Early Pancreas Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Virginia Mason Hospital/Medical Center (Other); VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0335-18-FB; U01CA210240-06 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes; Pancreas Cyst; Chronic Pancreatitis; Genetic Predisposition to Disease; Inherited Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Pancreatic Cyst; Pancreatitis, Chronic; Genetic Predisposition to Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Detection of early PDAC will ideally use clinical and/or biochemical markers of early disease in combination with novel imaging techniques to identify disease much earlier than current modalities. This study will focus on clinical symptoms and blood biomarkers and will allow the study of novel biomarkers in development using banked blood specimens. Identifying individuals with new-onset diabetes and/or diabetes in the setting of chronic pancreatitis, and who have clear evidence of type 3c diabetes may allow for targeted screening of these individuals, with Mixed Meal Tolerance Test, for pancreas cancer in light of the high risk of cancer in these individuals.
  Blood may be analyzed for other markers which are currently in development. NOTE: Blood must be collected in Omaha.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- New Onset Diabetes/High-Risk Prediabetes: Must meet one of the following criteria:
  1. New onset type 2 diabetes diagnosed within the past 3 years, defined as Hemoglobin A1c ≥ 6.5%*, fasting blood glucose >126mg/dL confirmed on a subsequent day or as diagnosed by a physician
  2. High-risk pre-diabetes: Hemoglobin A1c >6.3% or A1c >6.0% with fasting blood glucose >110 or 2 hour oral glucose tolerance test between 140-200mg/dL; subjects who have been on metformin <3 years are eligible
- Pancreatic Cystic Neoplasm/Pancreatitis: Must meet one of the following criteria:
  1. Pancreatic cystic neoplasm for which resection, endoscopic ultrasound or serial imaging has been recommended
  2. Chronic pancreatitis as defined by cross-sectional imaging, endoscopic ultrasound, functional testing abnormalities OR as diagnosed by a gastroenterologist
- Inherited Risk: Must meet one of the following criteria:
  1. Two or more blood relatives with PDAC (includes 1st-3rd degree relatives as defined in Table 2)
  2. One 1st degree relative with PDAC diagnosed before age 60
  3. Germline mutation associated with a higher than average risk of PDAC including but not limited to the following: Hereditary breast and ovarian cancer syndromes BRCA1, BRCA2, PALB2 Hereditary nonpolyposis colon cancer (Lynch) syndrome MLH1, MSH2, MSH6, PMS2 Familial adenomatous polyposis (APC) Familial atypical multiple melanoma and mole syndrome CKDN2a, p16 Peutz-Jeghers syndrome STK11 Ataxia-telangiectasia ATM Juvenile polyposis syndromes SMAD4, BMPR1A Li Fraumeni TP53 Cystic fibrosis and unaffected carriers CFTR
  4. Personal or family history which meets clinical criteria for a hereditary cancer syndrome and includes a relative with PDAC

SUMMARY:
Identifying biomarkers of early pancreatic ductal adenocarcinoma (PDAC) could facilitate screening for individuals at higher than average risk and expedite the diagnosis in individuals with symptoms and substantially improve an individual's chance of surviving the disease.

The investigators propose a longitudinal study of subjects at higher than average risk of PDAC in order to generate clinical data and bank serial blood specimens.

DETAILED DESCRIPTION:
Patients diagnosed with pancreatic ductal adenocarcinoma (PDAC) have only an 10% chance of surviving 5 years after diagnosis. Most PDAC is advanced and not amenable to curative therapies at the time of diagnosis, owing to lack of symptoms in early disease, nonspecific symptoms when they do develop resulting in a delay in diagnosis. Identifying biomarkers of early PDAC could facilitate screening for individuals at higher than average risk and expedite the diagnosis in individuals with symptoms and substantially improve an individual's chance of surviving the disease.

The investigators propose a longitudinal study of participants at higher than average risk of PDAC in order to generate clinical data and bank serial blood specimens. Participants will include individuals with family history of pancreas cancer, individuals with cystic pancreas lesions or chronic pancreatitis, and individuals with new-onset diabetes. Identifying specific biomarkers - blood markers and/or a clinical "prodrome" - in participants who go on to develop PDAC could improve the diagnostic approach outcomes for patients diagnosed with PDAC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19
* Able to provide written, informed consent
* Able to attend an in-person study visit in Omaha, NE twice a year to collect blood samples
* Must also meet criteria for one specific cohort. Participants who meet criteria for more than one cohort are eligible. (The intent being that potential participants must meet the criteria for at least one cohort, but are eligible if criteria are met for more than one cohort)

  o New onset diabetes/high-risk pre-diabetes cohort: must meet one of the following criteria: New onset type 2 diabetes diagnosed within the past 3 years, defined as A1c ≥ 6.5%, fasting blood glucose >126mg/dL confirmed on a subsequent day or as diagnosed by a physician High-risk pre-diabetes: A1c >6.3% or A1c >6.0% with fasting blood glucose >110 or 2 hour oral glucose tolerance test between 140-200mg/dL, or taken metformin <3 years

  o Pancreatic cystic neoplasm/pancreatitis cohort: must have one of the following diagnoses: Pancreatic cystic neoplasm for which resection, endoscopic ultrasound (EUS) or serial imaging has been recommended Chronic pancreatitis as defined by cross-sectional imaging, endoscopic ultrasound, functional testing abnormalities OR as diagnosed by a gastroenterologist

  o Inherited risk cohort: must meet one of the following criteria: Two or more blood relatives with pancreatic ductal adenocarcinoma (PDAC), includes 1st-3rd degree relatives (First - parent, sibling or child; Second - grandparent, aunt/uncle, niece/nephew, or half-sibling; Third - first cousin, great grand parent or great grandchild) One 1st degree relative with PDAC diagnosed before age 60; Germline mutation associated with a higher than average risk of PDAC, including but not limited to: Hereditary breast and ovarian cancer syndromes (BRCA1, BRCA2, PALB2) Hereditary nonpolyposis colon cancer (Lynch) syndrome (MLH1, MSH2, MSH6, PMS2) Familial adenomatous polyposis (APC) Familial atypical multiple melanoma and mole syndrome (CKDN2a, p16) Peutz-Jeghers syndrome (STK11) Ataxia-telangectasia (ATM) Juvenile polyposis syndromes (SMAD4, BMPR1A) Li Fraumeni (TP53) Cystic fibrosis and unaffected carriers (CFTR) Personal or family history which meets clinical criteria for a hereditary cancer syndrome and includes a relative with PDAC (as above)

Exclusion Criteria:

* Personal history of pancreatic ductal adenocarcinoma (PDAC)
* Currently receiving treatment for a cancer diagnosis (excluding long-term hormonal therapy)
* Pre-diabetes on metformin for ≥ 3 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In order to obtain a resource of clinical data and longitudinally obtained, annotated blood specimens and to develop an enriched population to prospectively evaluate a sensitive and specific biomarker, subjects from the following 3 groups at higher than average risk of pancreatic ductal adenocarcinoma (PDAC) will be recruited and enrolled.
  New onset diabetes, high risk pre-diabetes Pancreatic cystic neoplasms and pancreatitis Familial risk
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of pancreas cancer cases diagnosed. | 10 years
  Number of pancreas cancer cases diagnosed.
Biomarkers which may predict early pancreas cancer. | 10 years
  Biomarkers which may predict early pancreas cancer.
Result of MMTT which may indicate type 3c diabetes, which may be a risk factor for pancreas cancer. | 10 years
  Result of MMTT which may indicate type 3c diabetes, which may be a risk factor

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey A Klute, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The Pancreatic Cancer Detection Consortium (PCDC) includes collaborators at several institutions, including UNMC, working to identify biomarkers and develop novel imaging techniques to identify pre-malignant and subclinical PDAC. One of the primary objectives of the consortium is to establish a repository of serial biospecimens collected from subjects prior to their diagnosis of PDAC. These specimens will be readily available when biomarkers in development are ready for validation. Due to the low incidence of pancreas cancer, even in groups at substantially increased risk, obtaining enough specimens to use for biomarker identification from those subjects who go on to develop PDAC requires collaborative effort between multiple institutions. This proposal is the contribution from UNMC to the consortium's biorepository effort.
Time Frame: Data will be shared with the consortium on a rolling basis throughout the enrollment period.
Access Criteria: Priority will be given to researchers affiliated with the PCDC. Primary investigators will review outside requests, which may be accepted on a case by case basis.